





# Guided Self Help Following Sexual Assault

4 WEEKLY SESSIONS SCRIPTS & HANDOUTS

## Contents

| Seript | Session 1 – Introduction & Psychoeducation | 3 |
|---|---|---|
| Aims of session 1 66 Mindful Breathing Exercise 68 Reflection: What would you like from your sex life? 6 How difficult experiences get in the way 6 The brains alarm system 7 Reflection: What makes sex enjoyable for you? 7 Sex & Emotions: Three Systems 8 A Compassionate Approach 9 Week I Practice: 9 Session 2 - Being in the present moment and Grounding techniques 10 Seript 10 Session 2: Handout 15 Living Everyday on Autopilot 15 What is Mindfulness? 15 How can mindfulness and being present help after trauma? 16 Everyday Mindfulness 6 Practice: being present with mindfulness 16 Managing flashbacks during sex 17 54321 Grounding 17 Week 2 Practice: 18 Sesion 3 - Desire and the sensual self 19 Script 19 Script 23 Desire in Relationship 23 Inner S | <u>Script</u> | 3 |
| Reflection: What would you like from your sex life? 6 How difficult experiences get in the way. 6 The brains alarm system. 7 Reflection: What makes sex enjoyable for you? 7 Sex & Emotions: Three Systems 8 Three Systems after Trainna 8 A Compassionate Approach 9 Week 1 Practice: 9 Session 2 – Being in the present moment and Grounding techniques 10 Seript 10 Session 2: Handout 15 Living Everyday on Autopilot 15 What is Mindfulness? 15 How can mindfulness and being present help after trauma? 16 Everyday Mindfulness 16 Practice: being present with mindfulness 16 Managing flashbacks during sex 17 4321 Grounding 17 Week 2 Practice: 18 Sesion 3 – Desire and the sensual self 19 Seript 23 Desire in Relationship 23 Inner Sex Critic 24 Compassionate Self Exercise 25 <t< th=""><th>Aims of session 1</th><th>6</th></t<> | Aims of session 1 | 6 |
| Reflection: What makes sex enjoyable for you? 7 Sex & Emotions: Three Systems 8 Three Systems after Trauma. 8 A Compassionate Approach 9 Week I Practice: 9 Session 2 - Being in the present moment and Grounding techniques 10 Script 10 Session 2: Handout. 15 Living Everyday on Autopilot 15 What is Mindfulness? 15 How can mindfulness and being present help after trauma? 16 Everyday Mindfulness 16 Practice: being present with mindfulness 16 Managing flashbacks during sex 17 54321 Grounding 17 Week 2 Practice: 18 Sesion 3 - Desire and the sensual self 19 Script 23 Desire in Relationship 23 Inner Sex Critic 24 Compassionate Self Exercise 25 Activities to build on sensual self 25 Practice: Compassionate Letter Writing 25 Sesion 4 - Psychosexual techniques and relationships with others <t< td=""><td>Reflection: What would you like from your sex life?</td><td>6</td></t<> | Reflection: What would you like from your sex life? | 6 |
| Three Systems after Trauma 8 A Compassionate Approach 9 Weck 1 Practice: 9 Session 2 - Being in the present moment and Grounding techniques 10 Script 10 Session 2: Handout 15 Living Everyday on Autopilot 15 What is Mindfulness? 15 How can mindfulness and being present help after trauma? 16 Everyday Mindfulness 16 Practice: being present with mindfulness 16 Managing flashbacks during sex 17 4321 Grounding 17 Week 2 Practice: 18 Session 3 - Desire and the sensual self 19 Script 19 Serion 3: Handout 23 Re-learning Sex 23 Desire in Relationship 23 Locy of the compassionate Self Exercise 25 Activities to build on sensual self 25 Practice: Compassionate Letter Writing 25 Sesion 4 - Psychosexual techniques and relationships with others 26 Seript 26 <td< td=""><td>Reflection: What makes sex enjoyable for you?</td><td>7</td></td<> | Reflection: What makes sex enjoyable for you? | 7 |
| Sersion 2 - Being in the present moment and Grounding techniques 10 Script 10 Session 2: Handout. 15 Living Everyday on Autopilot 15 What is Mindfulness? 15 How can mindfulness and being present help after trauma? 16 Everyday Mindfulness 16 Practice: being present with mindfulness 16 Managing flashbacks during sex 17 4321 Grounding 17 Week 2 Practice: 18 Sesion 3 - Desire and the sensual self 19 Script 23 Desire in Relationship 23 Inner Sex Critic 24 Compassionate Self Exercise 25 Activities to build on sensual self 25 Practice: Compassionate Letter Writing 25 Session 4 - Psychosexual techniques and relationships with others 26 Seript 26 Session 4: Handout 30 Exercise: Compassionate Colour 30 Conditions for good sex 30 Relationships 31 Activ | <u>Three Systems after Trauma</u> . <u>A Compassionate Approach</u> | 8<br>9 |
| Session 2: Handout. 15 Living Everyday on Autopilot 15 What is Mindfulness? 15 How can mindfulness and being present help after trauma? 16 Everyday Mindfulness 16 Practice: being present with mindfulness 16 Managing flashbacks during sex 17 54321 Grounding 17 Week 2 Practice: 18 Session 3 – Desire and the sensual self 19 Script 19 Session 3: Handout 23 Re-learning Sex 23 Desire in Relationship 23 Inner Sex Critic 24 Compassionate Self Exercise 25 Activities to build on sensual self 25 Practice: Compassionate Letter Writing 25 Sesion 4 – Psychosexual techniques and relationships with others 26 Seript 26 Session 4: Handout 30 Exercise: Compassionate Colour 30 Conditions for good sex 30 Relationships 30 Activities involving physical touch | Session 2 – Being in the present moment and Grounding techniques | 10 |
| Living Everyday on Autopilot 15 What is Mindfulness? 15 How can mindfulness and being present help after trauma? 16 Everyday Mindfulness 16 Practice: being present with mindfulness 16 Managing flashbacks during sex 17 54321 Grounding 17 Week 2 Practice: 18 Session 3 – Desire and the sensual self 19 Script 19 Session 3: Handout 23 Re-learning Sex 23 Desire in Relationship 23 Inner Sex Critic 24 Compassionate Self Exercise 25 Activities to build on sensual self 25 Practice: Compassionate Letter Writing 25 Session 4 – Psychosexual techniques and relationships with others 26 Session 4: Handout 30 Exercise: Compassionate Colour 30 Conditions for good sex 30 Relationships 30 Activities involving physical touch 31 Week 4 Practice: 31 Appendix 32 | | |
| Everyday Mindfulness 16 Practice: being present with mindfulness 16 Managing flashbacks during sex 17 54321 Grounding 17 Week 2 Practice: 18 Session 3 - Desire and the sensual self 19 Seript 19 Session 3: Handout 23 Re-learning Sex 23 Desire in Relationship 23 Inner Sex Critic 24 Compassionate Self Exercise 25 Activities to build on sensual self 25 Practice: Compassionate Letter Writing 25 Session 4 - Psychosexual techniques and relationships with others 26 Seript 26 Session 4: Handout 30 Exercise: Compassionate Colour 30 Conditions for good sex 30 Relationships 30 Activities involving physical touch 31 Week 4 Practice: 31 Appendix 32 | Living Everyday on Autopilot What is Mindfulness? | 15<br>15 |
| Managing flashbacks during sex 17 54321 Grounding 17 Week 2 Practice: 18 Session 3 – Desire and the sensual self 19 Script 19 Session 3: Handout 23 Re-learning Sex 23 Desire in Relationship 23 Inner Sex Critic 24 Compassionate Self Exercise 25 Activities to build on sensual self 25 Practice: Compassionate Letter Writing 25 Session 4 – Psychosexual techniques and relationships with others 26 Script 26 Session 4: Handout 30 Exercise: Compassionate Colour 30 Conditions for good sex 30 Relationships 30 Activities involving physical touch 31 Week 4 Practice: 31 Appendix 32 | Everyday Mindfulness | 16 |
| Session 3 - Desire and the sensual self 19 Script 19 Session 3: Handout 23 Re-learning Sex 23 Desire in Relationship 23 Inner Sex Critic 24 Compassionate Self Exercise 25 Activities to build on sensual self 25 Practice: Compassionate Letter Writing 25 Session 4 - Psychosexual techniques and relationships with others 26 Script 26 Session 4: Handout 30 Exercise: Compassionate Colour 30 Conditions for good sex 30 Relationships 30 Activities involving physical touch 31 Week 4 Practice: 31 Appendix 32 | Managing flashbacks during sex 54321 Grounding | 17<br>17 |
| Script 19 Session 3: Handout 23 Re-learning Sex 23 Desire in Relationship 23 Inner Sex Critic 24 Compassionate Self Exercise 25 Activities to build on sensual self 25 Practice: Compassionate Letter Writing 25 Session 4 - Psychosexual techniques and relationships with others 26 Seript 26 Session 4: Handout 30 Exercise: Compassionate Colour 30 Conditions for good sex 30 Relationships 30 Activities involving physical touch 31 Week 4 Practice: 31 Appendix 32 | | |
| Re-learning Sex23Desire in Relationship23Inner Sex Critic24Compassionate Self Exercise25Activities to build on sensual self25Practice: Compassionate Letter Writing25Session 4 - Psychosexual techniques and relationships with others26Script26Session 4: Handout30Exercise: Compassionate Colour30Conditions for good sex30Relationships30Activities involving physical touch31Week 4 Practice:31Appendix32 | | |
| Re-learning Sex23Desire in Relationship23Inner Sex Critic24Compassionate Self Exercise25Activities to build on sensual self25Practice: Compassionate Letter Writing25Session 4 - Psychosexual techniques and relationships with others26Script26Session 4: Handout30Exercise: Compassionate Colour30Conditions for good sex30Relationships30Activities involving physical touch31Week 4 Practice:31Appendix32 | <del></del> | |
| Compassionate Self Exercise25Activities to build on sensual self25Practice: Compassionate Letter Writing25Session 4 - Psychosexual techniques and relationships with others26Seript26Session 4: Handout30Exercise: Compassionate Colour30Conditions for good sex30Relationships30Activities involving physical touch31Week 4 Practice:31Appendix32 | Re-learning Sex. Desire in Relationship | 23<br>23 |
| Practice: Compassionate Letter Writing25Session 4 - Psychosexual techniques and relationships with others26Session 4: Handout30Exercise: Compassionate Colour30Conditions for good sex30Relationships30Activities involving physical touch31Week 4 Practice:31Appendix32 | Compassionate Self Exercise | 25 |
| Script 26 Session 4: Handout 30 Exercise: Compassionate Colour 30 Conditions for good sex 30 Relationships 30 Activities involving physical touch 31 Week 4 Practice: 31 Appendix 32 | | |
| Session 4: Handout 30 Exercise: Compassionate Colour 30 Conditions for good sex 30 Relationships 30 Activities involving physical touch 31 Week 4 Practice: 31 Appendix 32 | <u>Session 4 – Psychosexual techniques and relationships with others</u> | 26 |
| Exercise: Compassionate Colour30Conditions for good sex30Relationships30Activities involving physical touch31Week 4 Practice:31Appendix32 | <u>Script</u> | 26 |
| Relationships30Activities involving physical touch31Week 4 Practice:31Appendix32 | Exercise: Compassionate Colour | 30 |
| Appendix | Relationships Activities involving physical touch | 30<br>31 |
| | Appendix | 32 |

## **Session 1 – Introduction & Psychoeducation**

## **Script**

#### Introduction:

Hello and welcome to the first session of guided self-help for sexual distress. Over the next 4 sessions we hope to cultivate a more compassionate view towards yourself by deepening your understanding of yourself and your difficulties, and how your experience of sexual trauma is affecting your sex life and the it affects your mind and body.

We have based this information from scientific research and throughout the sessions, we will also be going through a range of exercises for you to practice and ask for you to note down any reflections you feel comfortable writing. You have the choice of which exercises you want to try and which you would prefer to opt out of. It is completely okay to step away from any of the exercises over the next 4 weeks, you do what feels right for you. Even choosing to sign up for this 4 week intervention is a big step and we hope that this guide will help you feel more confident in returning to sex and treat yourself with more kindness when approaching sex even if it feels like it may be difficult.

#### Breathing exercise:

Breathing is a great form of mindfulness which cultivates our ability to be present in the moment. We will learn more about mindfulness in the next session. To help you prepare for today's session I would like to bring you to the present moment, let's get into a comfortable position and start by taking a deep breathe and relaxing any tension you may feel in your body. Take yourself away from any distractions and if you feel comfortable to do so. you can close your eyes and take a minute or two to allow your attention to settle on your breathing – not really thinking about anything in particular. Alternatively, or when you are ready, take one last deep breathe, stretch wiggle your finger and toes and bring yourself back in to the room.

#### Reflection:

To begin the session, I would like you to think about how you want to feel about your sex life and what about sex is important to you. Is it pleasure? Connection? Is not important to you. Take as much time as you need to reflect on this. If how you want to feel about your sex life is a 10 on a scale of 0 to 10, how close are you to feeling the way you want about your sex life?. What number would you rate your sex life currently from 0 to 10.

## How difficult experiences get in the way:

Research has shown how it is common and understandable for sexual trauma to affect someone's experiences of sex. For some people this changes the way they have sex or can lead to increased anxiety & fear of having sex and discomfort during sex. On the handout are a list of common experiences survivors of sexual trauma encounter when returning to sex. These experiences are understandable after trauma which is a violation of your safety and this is the way your brain is trying to protect you from being hurt again but it overcompensates, causing these symptoms. If you have any of these experiences currently, it is not your fault! You did not choose or want to react in these ways but our brains automatic response is to keep you safe.

The main task of all living things is survival and humans have evolved in many ways to detect and respond to threat to ensure we survive. The brain has also evolved to detect threat. The amygdala is the part of the brain that protects us from threat – it is the human built in threat alarm system. To protect us, the amygdala is constantly looking out for threat and lives by the rule 'better safe than sorry' so any small signs of danger can cause the alarm system to go off and our brain is told that we are in danger and prepares our body and mind to defend itself. This response occurs so quickly and automatically that sometimes it sets off our threat system before we are conscious of what is happening.

For example, if we are in a forest and see something moving on the ground we might feel scared and jump back before we realise it's a harmless bird. The role of the amygdala is to keep us safe and to react quickly before the thinking part of our brain identifies the movement as something that isn't dangerous.

Unfortunately, the amygdala is unable to distinguish between danger in the present from past events we remember in our minds. This is why the threat system may be activated when you have memories of trauma even if you rationally know you are in a safe place. Your brains is trying to keep you safe and prevent anything frightening from happening again. During the trauma, the amygdala collects information so that it can recognise warning signs in the future to prevent the event from occurring again. Anything that even vaguely reminds the amygdala of the original traumatic event, including the act of sex in a safe place on your own or with a trusted partner can trigger the threat system, When the 'alarm system' goes off because our threat system is triggered, it can interfere with the ability to have sex. I hope you will be reassured that many of the difficulties you experience are the results of the way the human brain is designed and to deal with threat.

The way our bodies respond sexually is related to a whole range of factors, many of which are outside our control such as the response of the threat system. One thing we can do to reduce the emphasis on the threat system is to activate our soothing system.

The soothing system is part of the three systems model and is linked to feelings of being safe and soothed. It is associated with being relaxed, connecting to others and experiencing compassion. Often for sex to be enjoyable we need: human connection, feeling safe, feeling wanted and our wishes respected. And a feeling of safety and no active threat. – these are all factors associated with the soothing system which is needed for arousal and enjoyable sex.

#### Three Systems:

We have already introduced how the threat system can interfere during sex. We also briefly talked about how the soothing system is what makes us feel safe during sex allowing for arousal. These two systems, described above, are part of a three systems model. The third system is the drive system and it's involved in wanting and pursuing sex. From an evolutionary perspective, the principle aim of sex is reproduction. However, we know that is not everybody's drive for sex today.

After experiencing trauma, the threat system becomes more sensitive and is easily triggered, overruling the drive and soothing systems as your brain tries to protect you from being hurt again even if you are with a trusted partner. This may cause people to feel:

- → unsafe, scared of sex etc.
- → shame about what happened, disgusted with self or others.

- → Some people worry that what happened to them was their fault, so might feel shame and feel undeserving of sex or closeness
- → Might have critical thoughts like "I'm disgusting" or "I'm not worth it"

Our brains and bodies are not designed to have sex "perfectly" (e.g. in the way our **culture** currently says we should) ... we're evolved to survive...

It is understandable that if someone has had a threatening or unwanted sexual experience, sex might be experienced as threatening. A new sexual encounter might automatically trigger memories of the unwanted sexual experience **OR** sex drive might increase — as the brain's way of managing the increased threat. This can be **automatic and unconscious**, and happen even if the person doesn't want it to. The brain is doing what it thinks is helpful, even if it doesn't feel helpful.

#### Building Compassion:

Over the next few weeks, we will work on acknowledging the difficulties and shame related to sex while building on the soothing system through different exercises. Increasing our soothing system will help increase our drive and alleviate the threat system. We do this by trying to be more compassion with ourselves. This includes

- → Understanding the way, we are and why we may act/feel this way being wise about sex and our bodies
- → Treating ourselves with warmth and kindness
- → Being encouraging to ourselves
- → Being non-judgmental about our experiences

Being compassionate will also allow us to be aware and engage with distress and difficulty without turning away from it and increase our motivation and courage to try to alleviate the distress.

#### Practice:

At the bottom of your handout there are some practice activities we encourage you to try throughout the week. It is perfectly okay to do all of them, some of them or none of them as long as you are doing what feels right for you. There is no pressure or need to be harsh with yourself if you were unable to incorporate these practices during the week, you are doing the best you can and being here for this first session is enough. Thank you for joining this week, this is a brief reminder to fill out the measures and questionnaires so that we can see how this intervention is helpful for survivors of sexual trauma. Thank you very much and I hope you found today's session helpful, we will see you next week.

## **Handout**

## Aims of session 1

- To think about what you'd like from your sex life
- To understand the links between difficult experiences and sex
- To understand why our brains and bodies act the way they do
- To build compassion towards the ways our minds and bodies behave

## Mindful Breathing Exercise

Reflection: How would you like to feel about your sex life?

## How difficult experiences get in the way

- Difficult / traumatic experiences can affect experiences of sex
- For some people, this can lead to anxiety, fear, discomfort around sex, or change the way you have sex
- This is <u>very understandable</u> as our brains are programmed to protect us and keep us safe it's not your fault!!!

# Listed below are common experiences survivors of sexual trauma have when returning to sex based on scientific research.

- → Decreased sexual satisfaction<sup>1</sup>,<sup>2</sup>
- $\rightarrow$  Decreased frequency of sex<sup>2,3</sup>
- $\rightarrow$  Fear of sex<sup>2</sup>
- → Difficulties with arousal/desire during sex<sup>2,4</sup>
- → Painful sex<sup>5</sup>
- → Lower sex drive
- → Higher sex drive<sup>5,6</sup>

- → Feelings of shame & self-blame<sup>6, 7</sup>
- → Avoidance of sex and/or connection <sup>1</sup>
- → Flashbacks<sup>1</sup>
- → Difficulties in trusting others<sup>6</sup>
- → Difficulties with relationships and communications<sup>6</sup>

These difficulties can be unpleasant but are understandable & expected responses to trauma. Having these experience does not mean you want or choose to have them –it is just the brain's automatic way of trying to protect us.

<sup>&</sup>lt;sup>1</sup> Norris, J., & Feldman-Summers, S. (1981). Factors related to the psychological impacts of rape on the victim. *Journal of Abnormal Psychology*, 90(6), 562.

<sup>&</sup>lt;sup>2</sup> Van Berlo, W., & Ensink, B. (2000). Problems with sexuality after sexual assault. *Annual review of sex research*, *11*(1), 235-257.

<sup>&</sup>lt;sup>3</sup>Feldman-Summers, S., Gordon, P. E., & Meagher, J. R. (1979). The impact of rape on sexual satisfaction. *Journal of Abnormal Psychology*, 88(1), 101

<sup>&</sup>lt;sup>4</sup>Becker, J. V., Skinner, L. J., Abel, G. G., Axelrod, R., & Cichon, J. (1984). Sexual problems of sexual assault survivors. *Women & Health*, *9*(4), 5-20.

<sup>&</sup>lt;sup>5</sup> Weaver, T. L. (2009). Impact of rape on female sexuality: Review of selected literature. Clinical Obstetrics and Gynecology, 52(4), 702-711.

<sup>&</sup>lt;sup>6</sup> O'Callaghan, E., Shepp, V., Ullman, S. E., & Kirkner, A. (2019). Navigating sex and sexuality after sexual assault: A qualitative study of survivors and informal support providers. The Journal of Sex Research, 56(8), 1045-1057.

<sup>&</sup>lt;sup>7</sup> Hamrick, L. A., & Owens, G. P. (2019). Exploring the mediating role of self-blame and coping in the relationships between selfcompassion and distress in females following the sexual assault. Journal of clinical psychology, 75(4), 766-779.

## The brains alarm system



The amygdala is the part of the brain that protects us from threat – think of it as the brains alarm system. It is constantly looking out for threat and lives by the rule 'better safe than sorry' so any small signs of danger can cause the alarm system to go off and our brain is told that we are in danger and prepares our body and mind to defend itself. This responds occurs so quickly and automatically that sometimes it sets off our threat system before we are conscious of what is happening.

When this alarm system goes off because our our ability to become aroused and enjoy sex.

system is triggered, it can interfere with

What we need is to activate our system. However, the way in which our bodies respond sexually is related to a whole range of factors – many of which are completely outside of our control.

SOOTHING

- → Human connection, feeling safe, feeling wanted and our wishes respected basic human needs related to the soothing system
- → A feeling of safety and no active threat

However, when you have experienced trauma, your body and brain tries to protect yourself from being hurt again even when are with a trusted partner.

## Sex & Emotions: Three Systems



We have already introduced how the threat system can interfere during sex. We also showed how the soothing system is what makes us feel safe during sex allowing for arousal, these two systems are part of the three systems model as seen above. The third system is the drive system and it's involved in wanting and pursuing sex. From an evolutionary perspective, the principle aim of sex is reproduction.

#### **Three Systems after Trauma**



After experiencing trauma, the threat system becomes more sensitive and is easily triggered, overruling the drive and soothing systems. This causes people to feel

- → unsafe, scared of sex etc.
- → shame about what happened, disgusted with self or others.
- → Some people worry that what happened to them was their fault, so might feel shame and feel undeserving of sex or closeness
- → Might have self-blaming
- → critical thoughts like "I'm disgusting" or "I'm not worth it"

 $\rightarrow$ 

Our brains and bodies are not designed to have sex "perfectly" (e.g. in the way our **culture** currently says we should) ... we're evolved to survive...

It is understandable that if someone has had a threatening or unwanted sexual experience, sex might be experienced as threatening

A new sexual encounter might automatically trigger memories of the unwanted sexual experience

,Sex drive might increase – as the brain's way of managing the increased threat - this can be an automatic process and happens even if the person does not want it to

The brain is doing what it thinks is helpful, even if it doesn't feel helpful

## A Compassionate Approach



Increasing our soothing system will help increase our drive and alleviate the threat system. We do this by trying to be more compassion with ourselves. This includes

- → Understanding the way, we are and why we may act/feel this way being wise about sex and our bodies
- → Treating ourselves with warmth and kindness
- → Being encouraging to ourselves
- → Being non-judgmental about our experiences

Being compassionate will also allow us to be aware and engage with distress & difficulty without turning away from it and increase our motivation and courage to try to alleviate the distress

## Week 1 Practice:

| How does the threat system get in the way of your sex life? |
|-------------------------------------------------------------|

Acknowledging these difficulties and the emotions such as anger/shame that come along with them is the first step in building the soothing system to allow yourself to let go of some of these difficult feelings.

## Session 2 – Being in the present moment and Grounding techniques

## Script

Hello and welcome to the second session. Today's session focuses on being in the present moment. These days we are so busy multitasking and doing many things that we may not be living our lives fully present. Additionally, we also know that the experience of trauma can make it even harder to be present because our minds may be elsewhere thinking about past events and at times, you may get involuntarily pulled into flashbacks or trauma memories without wanting to experience these memories.

In this session, we will learn about being present also known as mindfulness and learning about grounding techniques. As with each week, the core of these sessions is to build compassion towards the way our minds and bodies behave. We will practice some mindfulness exercises and I invite you to participate in whatever way feels right for you. With each exercise, you can choose if you want to try it and even if you choose not to, that's okay. You have showed up today and that can be enough.

#### Mindfulness - Living Everyday on Autopilot

We do many things every day without thinking or being aware of what we are doing. Think about times you are travel between two places and don't really remember the journey. Still, before you know it, you've arrived at your destination. **We call this autopilot mode**. In many ways, it can help us – routine tasks can be done easily, without thought. However, it also means we do many things without much awareness of what is happening and fail to be fully present and get the most from the experience. Living in autopilot also means our minds are less focused on what we are doing, and instead, it may be elsewhere. If you've had an experience of sexual assault, your mind may wander onto things associated with that experience even when you are doing something completely different. However, it is also common to think about the past experience of sexual assault when you are intimate with a partner. In the same way a task such as making a cup of tea becomes an automatic habit, so can worrying thoughts, unhelpful behaviours, and difficult feelings become an automatic habit if we are not conscious of being in the present.

Mindfulness offers a way to step out of autopilot and the unhelpful habits that come with it. It can help us get more from our day to day experience – to be more present in the things that we do. But it can also allow us to step back from difficult emotions – to be less caught up in them.

Mindfulness can be described as: <u>awareness</u> of <u>present moment</u>with <u>acceptance</u>. So, what do we mean by this? If we take each of the three phrases underlined above in turn, we can understand this statement better.

Awareness can be broken down into three steps:

#### Stop or slow down

When we are acting in autopilot we respond to situations, thoughts and emotions in automatic ways. The first step towards being more mindful, is to stop or slow down what you were doing – give yourself some space. Giving yourself some space can allow your mind to settle and provides a basis for reacting in a different way.

#### Observe

The next step is to observe what is going on for us. To do this, we first focus our attention on something - this can be on anything - e.g. and object around us, sounds that are going on around us. Most commonly, we can focus our attention on our breath. As we do so, we begin to notice the things that take our attention away from our breath. We notice where our attention goes.

#### Return

Once we have noticed that we have become distracted, that something has taken our attention away from our breath, we can note what has taken our attention away, and then return our attention back to our breath.

#### Present Moment

Sometimes we can be completely absorbed in the activity we are doing. However sometimes many things can take our attention away from our present experience. Mindfulness is a way to bring us back to the present moment.

#### Acceptance

The present moment is affected by how we view or judge it. To accept the present is to experience it without judging it. It is to see things in the moment as they are, not as we might want or expect them to be, or what we fear they might become. We are accepting our experience, pleasant or unpleasant, as it is.

## How can mindfulness help after trauma?

Studies have found that mindfulness helps reduce distracting thoughts, increases focus on physical sensation, and is helpful for sexual difficulties. It helps us learn to be in the moment by being aware of our physical sensations. And we want to build on compassion and activate our soothing system which we can do through mindfulness.

However, some survivors of sexual trauma may find mindfulness difficult or triggering and dissociates. Mindfulness may be quite distressing if it means sitting with sensations and emotions that are usually avoided. and If your mind 'shuts off' during your experience of trauma, the feeling of 'shutting off' can occur again when you're faced with similar or difficult emotions. If you experience these difficulties, it's okay. It's a protective mechanism to keep you safe. You can opt-out of the mindfulness exercise and practice being present in a different way. One way to do this is through everyday mindfulness.

#### **Everyday Mindfulness**

In any task we do, we can be mindful and present. Choose a routine task and each day for the next week; see if you can remember to pay attention while doing it. You do not have to slow it down or even enjoy it. Simply do what you normally do, but see if you can be fully alive to it as you do so.

Examples like: Brushing your teeth. Drinking a hot drink.

We are going to now have a short mindfulness practice – if you know mindfulness is difficult for you because of your experience of sexual trauma, you can skip the practice and I invite you

to do anything you find soothing or if you feel up for it, practice one of the everyday mindfulness activities instead. However, if you would like to give the activity a go, then continue and remember you have control and can stop and move on from this exercise at any point.

To begin, find a comfortable sitting position and if you feel comfortable, closing your eyes.

Mindfulness Attention Practice – based on Paul Gilbert's exercise. From Compassionate-Mind Guide to Recovering from Trauma and PTSD Deborah A. Lee

"Sit quietly for a moment and focus on your breathing. Allow the breath to come down into your diaphragm slowly and evenly and then leave your body slowly and evenly. If you find this difficult you may simply want to try to focus on the sensation of your breath coming in and leaving through your nose. Try spending two minutes simply concentrating on the experience of breathing in and out. If you don't like focusing on your breathing or you don't like closing your eyes, you could use a pebble or a shell and try to focus your attention on the experience of looking at it and feeling it or look at a blank wall.

As you focus on your in breath and out breath You may notice that within just a few moments your mind will have wandered off on to something else. This is called mind wandering. If there are things that are worrying us, our minds easily get pulled into thinking about them and away from the present moment. This can also happen if there are things we are looking forward to (like a party), or if there are things that we need to do (e.g., pay a bill, or remember to call a friend), and we can find our minds skipping to them. This is very typical of how our minds are, and indeed recent research evidence suggests that it is our natural state.

One aspect of practicing mindfulness is just learning to notice when our minds wander and bringing our attention gently and warmly back to what we want to focus on. Mindfulness is not making our minds pay attention or emptying our mind of thoughts. Telling ourselves off for not being able to pay attention is not being mindful either. Indeed, it is counterproductive, as noticing where our minds wander to can be very important in helping us to identify other issues that are bothering us. When our minds wander it is not a sign that we have failed to be mindful; it is a part of the very process of being mindful! It is the act of noticing and then returning the attention to the desired focus that is central to mindfulness. The very fact that you find this difficult is itself evidence that you are engaging in mindful practice!"

We are about to draw this mindfulness practice to a close so just focusing on you breathe for a few more moments and then feeling the weight of your body on the chair or floor and when you are ready, bringing yourself back into the room and open your eyes.

Before we move on I just want you to notice how you feel after that practice, you may feel relaxed, you may feel more tense or you may have noticed how you're not use to being present and your mind continued to wander. It's normal if this happens – Mindfulness is like a muscle and the more you practice the easier it gets. If you found the practice difficult as it triggered difficult feelings, you did your best to try out the exercise and should feel proud for being brave to do so. Instead of doing the mindfulness practice in future sessions, you can opt to do whatever you feel comfortable doing.

To finish the session today we will think about managing flashbacks during sex and grounding techniques you can use. Flashbacks are very common In any traumatic experience. And when you are a survivor sexual trauma, it is common for women to avoid sex because of the associations it brings up and the feelings, sensations and memories sex can trigger. It can be challenging to return to sex even if you are on your own or with a trusted partner. This is not because you chose or want to relive your past but experiencing flashbacks is understandably challenging and scary – it is not your fault that you experience them.

To manage flashbacks during sex, it can be helpful to have a conversation with your partner when you're not having sex. You can discuss why flashbacks occur and that they are not because of anything your partner has done wrong. You can also share or discuss the knowledge you've gained from this intervention with your partner. Remind your partner the confusion is not about them – it's about the situation. We know these conversations can be difficult – we have included a short brief handout (appendix B in your handout sheets) that you could share with your partner if you find it difficult to discuss your traumatic experience and your level of comfort during sex (Appendix B).

During this talk you can discuss with your partner the level of comfort with sex – are there any dos or don'ts specific to you? Anything you would prefer your partner to do/not do? This can start very simple e.g. holding hands, dancing, cuddling up in bed with a film. It can then branch into sexual things you feel comfortable with. We have included a sexual activities list and body map in your handout (Appendix C/D) to introduce the conversation. There is no pressure to do anything you are not comfortable doing, it's okay if this conversation takes time.

If you have been with the same partner prior to experiencing trauma, you may feel bad about having to change the way you have sex but it is not your fault. It may be more uncomfortable having these conversations with a casual partner but it's an important one to have to ensure you feel safe and more confident.

Du ring the discussion, you can plan of action with your partner with the aim to activate your soothing system. The plan can include

- Signal that flashback is occurring (e.g. specific arm pat, or word)
- An Okay to pause and take some time
- Might need to express emotion e.g. cry
- Use grounding technique (next slide)
- As part of grounding discuss with partner in advance how you would like them to respond in this situation. E.g. you might like partner to say, "it's okay, you are safe with me, I will not hurt you." You might like them to hold you while you feel sad, or for them to sit and listen to how you feel.
  - Breathe

This might occur a few times in sex before gradually over time you feel more comfortable and safe. Requires patience and compassion, both self-to-self and other-to-self.

If you have found things that have worked you can use those, these are only some ideas, you might have different ideas

Grounding Techniques are used to remind you where you are and that you are safe. It can be really helpful to discuss possible grounding techniques you can use with a sexual partner and communicate that with them. It can also be helpful to reflect on what you can use on your own. When thinking of grounding techniques, think about all 5 senses and how you can use your touch, smell, taste, sight and sound. You can write you own ideas below.

- Grounding object
- Sexual grounding object
- A phrase or object that reminds you WHERE you are and that you are SAFE. E.g. Item of clothing, a particular object (e.g. a stress ball, a ring, a special item) Or a piece of paper with the phrase "you are at your home, you are not in danger, you are safe".
- Using 5 senses for grounding
  - o Smell: essential oils. Candles
  - o Taste: mint/gum/sour candy
  - o Touch: weighted blanket, furry objects
  - O You can also use the 54321-grounding technique included in your handout the 54321-grounding technique is simple, yet powerful. Like gradually attaching anchors to the boat, this method slowly pulls you back to earth. It involves you naming 5 things you can see, 4 things you can touch, 3 things you can hear, 2 things you can smell and 1 thing you can taste.

With everything, there is no need to blame or be critical of yourself if you have to make a plan to be intimate and feel safe. Your threat system may activate when you are trying to have sex alone or with a partner because of your experience of trauma and that is not because you want or choose to have sexual distress – it's how our brains have evolved and are hardwired. It may also be uncomfortable to have these conversations with a partner, and that's understandable. It may be difficult to find the right words, feelings of shame or guilt, and some people may feel very vulnerable talking about this to anyone. If you experience any of this, it's not your fault. You have the power to choose when you are ready to have these conversations.

Practicing being present and having a plan should your threat system activate are ways we try to activate the soothe system to help you feel prepared and more confident in returning to sex.

#### Week 2 Practice:

- 1. Practise everyday mindfulness/ grounding technique choose one task to focus on for the whole week.
- 2. Listen to mindfulness audio every day to practice being in the present moment

**Session 2: Handout** 

## <u>Living Everyday on Autopilot</u>

We do many things every day without thinking or being aware of what we are doing. Think about times you are travelling between two places and you don't really remember the journey but before you know it, you've arrived at your destination. **We call this autopilot mode**. In many ways it can help us – routine tasks can be done easily, without thought. However, it also means we end up doing many things without much awareness of what is happening and fail to be fully present and getting the most from the experience. Living in autopilot also means our minds are less focused on what we are doing and instead it may be elsewhere. If you have an experience of sexual assault, your mind may often wander onto things associated with that experience even when you may be doing something completely different. However, it is also common to think about the past experience of sexual assault when you are intimate with yourself or a partner.

Mindfulness offers a way step out of autopilot and the unhelpful habits that come with it. It can help us to get more from our day to day experience – to be more present in the things that we do. But it can also help us to step back from difficult emotions – to be less caught up in them.

#### What is Mindfulness?

Mindfulness: <u>awareness</u> of <u>present experience</u> with <u>acceptance</u>. It's intentional, accepting and non-judgmental focus of one's attention on the present moment

#### **Awareness**

#### 1. Stop or slow down

When we are acting in autopilot we respond to situations, thoughts and emotions in automatic ways. The first step towards being more mindful, is to stop or slow down what you were doing – give yourself some space. Giving yourself some space can allow your mind to settle and provides a basis for reacting in a different way.

#### 2. Observe

The next step is to observe what is going on for us. To do this, we first focus our attention on something - this can be on anything - e.g. and object around us, sounds that are going on around us. Most commonly, we can focus our attention on our breath. As we do so, we begin to notice the things that take our attention away from our breath. We notice where our attention goes.

#### 3. Return

Once we have noticed that we have become distracted, that something has taken our attention away from our breath, we can note what has taken our attention away, and then return our attention back to our breath.

#### **Present Moment**

Sometimes we can be completely absorbed in the activity we are doing. However sometimes many things can take our attention away from our present experience. Mindfulness is a way to bring us back to the present moment.

#### **Acceptance**

The present moment is affected by how we view or judge it. To accept the present is to experience it without judging it. It is to see things in the moment as they are, not as we might want or expect them to be, or what we fear they might become. We are accepting our experience, pleasant or unpleasant, as it is.

## How can mindfulness and being present help after trauma?

Studies have found that mindfulness helps reduce distracting thoughts and increase focus on physical sensation and is helpful for sexual difficulties. It helps us learn to be in the moment by being aware of our physical sensations. Research has also shown that regular mindfulness practice increases genital response and psychological arousal.

However, we also know it can be really difficult for survivors of sexual trauma to practice mindfulness and may make you feel more disconnected or cause you to dissociate. This is understandable as your brain is trying to protect you from experiencing difficult emotions. If you are struggling to practice mindfulness that's okay. You can do other practices to be present!

## **Everyday Mindfulness**

Choose a routine task and, each day for the next week; see if you can remember to pay attention while you are doing it. You do not have to slow it down or even enjoy it.

Examples of routine tasks:

- Brushing your teeth
- Drinking tea, coffee, juice
- Walking to the shops
- Having a shower
- ..... (your choice!)

## Practice: being present with mindfulness

| eflection: How was that? |
|--------------------------|

## Managing flashbacks during sex

Have a conversation with a partner or reflect on your own abour flashback

Agree on safe and unsafe behaviours during sex Make a plan of action to deal with a flashback

Example actions to include

- Using specific grounding techniques
- A signal to inform your partner that you're having a flashback or want to stop
- Agreeing to pause if things begin to be difficult
- Acknowledging difficult emotions (e.g. fear/anger/disgust/shame)
- Breathing together and engaging soothing system

Grounding Techniques are used to remind you where you are and that you are safe. It can be really helpful to discuss possible grounding techniques you can use with a sexual partner and communicate that with them. It can also be helpful to reflect on what you can use on your own. When thinking of grounding techniques, think about all 5 senses and how you can use your touch, smell, taste, sight and sound. You can write you own ideas below.

## 54321 Grounding

Take a moment and take a few deep breaths invite your body back into the moment, slowing everything down. Then, become aware of your environment.

- Look For 5 Things You Can See: Notice the wood grain on the desk in front of you.
   Or the precise shape of your fingernails. Become aware of the glossy green of the plant in the corner. Take your time to really *look* and acknowledge what you see.
- Become Aware Of 4 Things You Can Touch: The satisfyingly rough texture of the
  car seat. Your cotton shirt against your neck. If you like, spend a moment literally
  touching these things. Maybe notice the sensation of gravity itself, or the floor beneath
  you.
- Acknowledge 3 Things You Can Hear: Don't judge, just hear. The distant traffic.

  The voices in the next room. As well as the space between sounds.

- Notice 2 Things You Can Smell: If at first you don't feel like you can smell anything, simply try to sense the subtle fragrance of the air around you, or of your own skin.
- **Become Aware Of 1 Thing You Can Taste:** The lingering suggestion of coffee on your tongue, maybe?

Repeat this process as many times as necessary. Take your time and notice how you feel afterward.



With everything, there is no need to blame or be critical toward yourself if you have to make a plan in order to be intimate and feel safe. Your threat system may activate when you are trying to have sex alone or with a partner because of your experience of trauma and that is not because you want or choose to have sexual distress – it's the way our brains have evolved and are hardwired. Practicing mindfulness and having a plan ready should your threat system activate are ways we try to activate the soothe system to help you feel prepared and more confident in returning to sex.

#### Week 2 Practice:

- 3. Practise everyday mindfulness/ grounding technique choose one task to focus on for the whole week.
- 4. Listen to mindfulness audio every day to practice being in the present moment

## <u>Session 3 – Desire and the sensual self</u>

## **Script**

Welcome to session 3. This week we will focusing on a very important relationship, the relationship you have with yourself.

To start the session, I would like you to reflect on all our beliefs about sex and how we learn about sex. If we start thinking about the natural behaviours we do as humans, such as walking and talking - these are things we naturally learnt to do. We needed a lot of support, coaching, guidance and patience from supportive caregivers to learn to walk. Even once we've learnt to walk, we might injure ourselves later in life (e.g. break a leg) and need to learn again. Recovery will be more effective with the help of compassion from others, patience and practice. Sex isn't any different to this – it's also something we learn. There's a myth that because sex is natural, we should instantly be 'good' at it. This isn't the case. Learning about what our bodies need and enjoy, and what our partners find pleasurable can take time. We might even have events later in life which set us back (e.g. infections/menopause/illness/child birth/trauma). Following this, sex might require re-learning and we might have to change our beliefs about sex. Sex is not static – sex is something that shifts and develops/changes over time and is something you can work on.

What are your beliefs about sex and where do they come from? Some example beliefs include

- Sex should always end in an orgasm
- If I'm in love, it should be easy
- Sex is only done in marriage
- Sex always involves vaginal penetration
- Everyone else is having great sex
- Sex should always be a deeply emotional experience OR the opposite, sex is only physical

These beliefs can come from family, culture, religion and societal norms. However, these beliefs can be unhelpful and make you feel worse about yourself. Many sexual difficulties result from one's own <u>assumptions and expectations</u> about sex. This is not because you are doing anything wrong, but we are taught to believe certain things about sex.

#### **Desire**

Similarly, we may have beliefs about desire arousal during sex.

Desire and arousal arise due to complex brain processes. Emily Nagoski is a sex educator and researcher, she explains how we can think of the processes that are involved in desire as a sexual accelerator that notices all sexually relevant information in your environment to turn you on BUT we also have the sexual brakes which notices all the reasons not to be turned on right now and neurologically tells your sexual system to turn off.

The process of being aroused is a two-way process of turning on the accelerator and turning off the brakes. Everyone accelerator and brakes have different sensitivities.

Difficulties with desire and arousal occurs if you cannot turn on the accelerator or more often, because there's too much stimulation on the brake.

Reflection: at this point it may be helpful to Reflect on what may turn on your sexual accelerator or what may cause your brakes to get stimulated – you may not have any answers and that's okay – there is not right or wrong answers here. It is just something that may be helpful for some of you to think about.

Unfortunately, the process gets more complex research has shown that if you are a stressed or in a threatened state of mind – your tricky brain will interpret almost any sensation as something to be avoided, as a potential threat and turn off the sexual accelerator while hitting hard on the sexual brakes. Telling your sexual system to turn off leading to reduced or no desire.

This is common for many individuals with or without an experience of sexual trauma and is not your fault. Some people may blame themselves for having increased or reduced desire after an experience of sexual assault but this is not something you have done to yourself. it's how your brain works to protect you even when it is unhelpful—The main goal of this intervention is not necessarily to increase desire or arousal for sex but to understand why you may be experiencing some of your difficulties and treat yourself more kindly since your challenges are not your fault. However, if you want to work on your desire, we have included some ideas in your hand out if you are ready to try.

#### Inner Sex Critic

One thing that does hit the brakes are self-blaming self- critical thoughts. It is a very common experience for survivors of sexual assault to have an inner sex critic who may be harsh and blaming towards yourself – this voice tells you things such as:

Why can't you do this?
There's something wrong with you
You'll never have a proper relationship
Everyone else finds sex easy
You'll never be able to enjoy sex
It's all pointless
You're weird
It's your fault
You don't deserve to have enjoyable sex?

The inner sex critic is part of the threat system, which is trying to protect you from getting hurt or experiencing trauma again. However ... it often does more damage than good. The inner sex critic can take different forms at different times. Sometimes it repeats what others have said or societal messages or expectations. Listening to the inner critic can be very painful and shouting at it to "shut up" doesn't usually work. It is one of the reasons we covered mindfulness as being present in the moment and how it helps you acknowledge the inner sex critic without buying into what they are saying.

Mindfulness gives us a way to acknowledge the inner sex critic without buying into what they are saying. It can also be helpful to think about what you may say to a friend if they experience the same difficulty. Would you tell them it's their fault they have sexual distress and weird that they can't do it? It is also helpful to develop an inner compassionate self to help you be kinder with yourself and build resilience to the inner sex critic.

We will now do a short exercise to develop your **compassionate self developed by Paul Gilbert**– as always if you do not feel comfortable doing this exercise, you can opt out before we begin and take some time now to do something nice for yourself. You also have the option to stop the exercise once we begin.

Get into a comfortable position and begin by focusing on your breathe. When you feel that your body has slowed down (even slightly) and you are ready for your practice, imagine that you are a very deeply compassionate person. Think of all the qualities that you would ideally have as that compassionate person. First focus on your desires to become a compassionate person and to be able to think, act and feel compassionately. Next, imagine being wise and having wisdom – a wisdom that comes from your understanding about the nature of our lives, of our minds and bodies and that there's so much that goes on inside of us which is not our fault but the result of evolution and experiences over which we had no control

Then when you are ready and have a sense of your wisdom, imagine having strength, maturity, authority. Explore your body posture – sit in a position in a way that matches your idea of being strong. Your facial expressions should also reflect your assertiveness and what it feels like to be confident. Remember you are imagining yourself as a person that understands one's difficulties and those of others, in a non-judgmental way, and has confidence to be sensitive, with an ability to tolerate difficulties.

When you are ready, move on to focusing on qualities of warmth and gentle friendliness. Imagine being warm and kind. Create a compassionate facial expression. Imagine yourself speaking to someone and hear the warm tone of your voice; imagine reaching out to someone with warmth and know what that might be like.

Then when you are ready switch to imagining a feeling of responsibility. Imagine that you have lost interest in condemning or blaming and are now wanting to do the best you can to help yourself and others move forward. Hold on to your compassion and facial expression of warmth, but just focus on this experience of taking up responsibility and committing yourself to being more compassionate with yourself.

Remember, it doesn't matter if you feel you have these qualities or not, just imagine that you have them. See in your mind yourself having them, and work through them steadily, playfully and slowly. Finally, imagine yourself having all of these qualities and incorporating them into the way you are with yourself and others.

When you have finished, bring yourself gently back into the room. You might want to write down what it felt like to have these qualities and how it might affect the way you want to act in the future.

If you like to take some time to write down how you feel after the exercise feel free to do so. Holding in mind your compassionate self, we would like to end the session thinking about your sensual self.

#### Sensual Self

Sexual trauma influences your sexual identity with a partner but more importantly, with yourself. When you have an experience of trauma it can trigger feelings of shame or guilt for feeling sexual or good about yourself. You may also let the needs of others overshadow your own needs and it is important to turn towards yourself by doing things every day for no one else's needs but your own.

Redefining your sexual self builds more ownership of your body, and helps you be in touch with your feelings and needs.

The sensual self is how you view sexually outside of relationships with other people. It can help build confidence in yourself and if you would like to return to sex, it can help increase desire and motivation for sex.

This could include wearing clothes that you enjoy, seeing someone on the street that you find attractive, moving your body in a way that feels good for you or wearing makeup that you love. Many of these things are part of the sexual self. These are also more gentle ways to explore your sexual self in small steps before considering being intimate with someone else. It may be helpful to think of rebuilding your sensual self as taking yourself on an adventure of learning more about yourself and what you enjoy.

Remember it takes time to rebuild your sensual self and learn to prioritise yourself after sexual trauma, so don't worry if this feels like a slow process, that's normal.

One way to work on the relationship with yourself and rebuild your sexual self is turning towards yourself with compassion and kindness. As a practice exercise for this week, I invite you to write yourself a compassionate letter. This letter is written by you and addressed to you.

The idea behind the compassionate letter comes from Paul Gilbert to help people engage with their difficulties with a focus on understanding and warmth towards themselves. It is to turn towards yourself in a non-judgemental way with a position of kindness and understanding of your difficulties instead of being harsh or blaming of yourself. (Appendix C). Towards the end of the compassionate letter you may also want to focus on being compassionate to your sensual self and consider how you can incorporate activities to build on yourself sensual self but what you decide to do is up to you,

We know it may not be easy to be compassionate with yourself and it is understandable if you find this exercise difficult. Not many people are used to being kind to themselves but we encourage you to try to do this exercise and see what happens over time. Research has also found that expressive writing can help people deal with difficult life experiences. When writing the letter, we encourage you to be empathetic and warm – as if you were writing to a loved one. Avoid going into 'I should or should not', 'why don't you' advice – be supportive and encouraging. We have included a guidance for this in this week's handout and encourage you to try the exercise sometime this week. However, if you are not able to now it's okay to opt out of the exercise. This letter will be your practice for this week, thank you for attending the session today, next week will be our final session.

## **Session 3: Handout**

| Re-learning Sex Reflection: What are your beliefs about sex? Where do they come from? |
|---|
| Desire in Relationship |
| brake accelerator or gas |
| Emily Nagoski simplifies the complex sexual processes that occur during arousal into two mechanisms – the sexual accelerator and the brakes. The accelerator and brakes are constantly seeking out information from everything you hear, see, touch, taste, smell and imagine. |
| • notices all the sexually relevant information in the environment and TURNS ON arousal |
| Sexual Brakes • notices all the relevant information and reasons not to be aroused and TURNS off arousal |
| The process of being aroused is a two-way process of turning on the sexual accelerator and stepping off the brakes. Difficulties with arousal mostly arise as there's too much stimulation to the brake and all kinds of things can hit the brake. |
| Reflection: What are the things that hit your sexual accelerator – TURN ON |
| What are the things that hits the brake – TURN OFF |

However, it's not just what the sexual accelerator and brake notices in your environment because research has shown that if you are a stressed out or in a threatened state of mind – your tricky brain will interpret almost any sensation as something to be avoided, as a potential threat and turn off the sexual accelerator while hitting hard on the sexual brakes.

#### Ideas to release the brake

- Begin with non-sexual touch either on your own or with a partner. There is no pressure for this touch to become sexual unless you feel comfortable for it to. Affection can signal to your brain that you are in a safe place and reduce stress.
- Create a stress free environment for yourself when you want to have sex on your own or with your partner—this can look like whatever you want lights on/off, having candles, calming music.
- Practice being present in the moment and focus on the sensations you feel currently
- Accepting yourself as you are and not being critical about what you are doing or how you look. This is much easier said than done but being self-blaming or listening to the inner self critic will hit the brakes.

#### Inner Sex Critic

Having an inner sex critic who criticises you is something that can step on the sexual brakes. If you experience an inner sex critic, this is not your fault, it is also really common for survivors of sexual assault to have an inner sex critic who tells you things such as:



The inner sex critic is part of the threat system which is trying to protect you from getting hurt or experiencing trauma again. However ... it often does more damage than good and can slam on the your brakes cause difficulties in desire and other areas of your sex life.

Mindfulness gives us a way to acknowledge the inner sex critic without buying into what they are saying. It can also be helpful to think about what you may say to a friend if they experience the same difficulty. Would you tell them it's their fault they have sexual distress and weird that they can't do it?

## Compassionate Self Exercise

| Reflection: |
|-------------|

## Activities to build on sensual self

Sexual trauma can change the way we view our selves sensually. Redefining your sensual self is an important step in gaining control over your body and becoming in tune with your emotional feelings. The sensual self is how you view sexually outside of relationships with other people/ It can help build confidence in yourself and if you would like to return to sex, it can help increase desire and motivation for sex.

- 1. Turning towards yourself with compassion
- 2. Doing things for yourself and not for others
  - → Wearing clothes you love
  - → Wearing make up that makes you feel confident
  - → Using products you like the feel of such as a nice moisturiser or hair mask
  - → Doing your hair in a way that you like
  - → Wearing jewellery that makes you feel good
  - → Getting a temporary tattoo that you like
- 3. Appreciating your body
  - → Moving your body in a way you like exercise, dancing, walking.
  - → Taking care of your body by stretching or pampering yourself with a face mask
  - → Giving yourself massages

## Practice: Compassionate Letter Writing

The idea behind the compassionate letter comes from Paul Gilbert to help people engage with their difficulties with a focus on understanding and warmth towards themselves. It is to turn towards yourself in a non-judgemental way with a position of kindness and understanding of your difficulties instead of being harsh or blaming of yourself.

#### Session 3 Practice Ideas

- 1. Listen back to the compassionate self audio throughout the week
- 2. Just as we discussed being mindful everyday, try to practice being compassionate with yourself daily
- 3. Gently explore your sensual self in any way that feels right for you
- 4. If you feel ready, write yourself a compassionate letter using the guidance provided in Appendix C

## Session 4 – Psychosexual techniques and relationships with others

## **Script**

Welcome to the final session. In the first session we covered your threat alarm system and how your body and brain tries to protect you after an experience of trauma. In the second session, we focused on being in the present moment through mindfulness and everyday mindfulness. We also covered grounding techniques which can be used to bring you back to the present moment. In the third session, we thought about the relationship you have with yourself and the tendency for people with experience of sexual trauma to develop a harsh inner critic. Throughout the last 3 sessions, we have woven in the idea of being kinder and more compassionate to yourself as a way to inhibit the threat system and trigger the soothing system. Being more understanding of yourself is an indirect way to aid in your confidence or motivation to return to sex. In our final session today, we will be introducing the conditions of good sex model and think more about your relationships with others as well as cover a range of psychosexual exercises that you can do alone or with a partner. As always, you have the choice to decide if you would like to try out these exercises. There is no pressure to do anything if you are not comfortable. We have included the links to handout for the exercises in the email instead of including it in this material so you have the choice to view them if you are interested and comfortable.

Let's begin with a short exercise and start by being compassionate with yourself as you have done so well to attend each week. As always, you can opt of this exercise and do something nice for yourself instead such as just taking a few deep breaths or preparing a nice warm or cool drink.

## Compassionate Colour Exercise - by Paul Gilbert

Sit in a comfortable position and if you feel comfortable, close your eyes. Beginning by focusing on your breath and when you're ready, imagine a colour that you associate with compassion, or a colour that conveys some sense of warmth and kindness. Again, it might only be a fleeting sense of colour but when you are ready, imagine your compassionate colour surrounding you. Then, imagine this entering through your heart area and slowly through your body. Or you might prefer to think of colour like a mist or light that just flows though you. As this happens try to focus on this colour as having wisdom, strength and warmth, with a key quality of total kindness. Create a facial expression of kindness on your own face as you do this exercise. Now, as you imagine the colour flowing through you focus on the feeling that the sole purpose of this colour is to help you, to strengthen you and support you.

To begin this session, we want to introduce this model of good sex. The conditions for good sex triangle consists of being in the moment, physical touch and psychological arousal. The conditions that you feel are important for psychological arousal and physical touch differ from person to person. Each condition also impacts each other. This triangle is a good way for you to reflect on your sex life currently. It can help you understand which area you may have more difficulties

In the last 4 weeks, we have covered being in the present moment and aspects of psychological arousal. Later we will think more about enjoying physical touch.



However, you can also see how communication with a sexual partner is an important condition and although we have briefly mentioned this in session 2 when we discussed grounding, we also want to think of how your relationship with others may change after sexual trauma.

#### Relationship with others

After traumatic sexual experiences, some people might notice a difference in their relationships or interactions with partner/s. – remember that this is not your doing but a common experience of anyone who has experienced trauma. Some partners may be understanding by responding with empathy and patience in relation to sexual intimacy

Others may struggle to understand, and could take a less helpful stance

If you are currently with a sexual partner/s, or would like to enter into a romantic or sexual relationship in the future, it can be helpful to reflect on the dynamics between you and your partner/s and consider the following:

→ How understood do you feel? How safe do you feel to engage in sex? How supportive is your partner of your needs and the pace you would like to take things? Are your 'conditions for enjoying sex and intimacy' being met?

If you find it difficult to be intimate with a partner, it may be helpful to first practice on your own

## Self-Practice – from sexualwellbeing for all

Mindful Self-Practice is A good way to feel more in tune with your own body and develop your sensuality is through exploring physical touch. One way to do this is through masturbation. I know it may be a awkward topic but self-practice is a great way to get to know your body, find out what you like but also helps you regain some control over your body. This can also feel like a safer first step before being intimate with a partner. Being mindful during self-practice means trying to focus on the physical sensations instead of allowing your mind to wander worrying about performance or self-criticism. If you are interested to try self-practice we have included a link to a more detailed handout by sexualwellbeingforall. If you are not comfortable with masturbation that's okay too, this can be about exploring touch in a way that feels safe for you and just getting to know your body.

 $\underline{https://sexualwellbeing for all.files.wordpress.com/2019/05/mindful-self-practice-forthose-with-a-vulva-1.pdf}$ 

#### Sensate Focus

If you have a trusted partner who you want to try an exercise with, you can try sensate focus which is practicing intimacy without genital contact. Sensate Focus is a set of exercises geared towards couples where the focus of sex is shifted from pursuing a particular outcome (e.g. penetration or orgasm), to a slower appreciation of physical intimacy and sensations. Sensate focus does not involve penetrative sex or other sex acts that can feel uncomfortable, painful or triggering, as the idea is to instead engage in various forms of giving and receiving touch that feel comfortable, unpressured and at a pace that feels right for you. Removing the pressure to achieve orgasm or have penetrative sex allows the partners to connect more deeply within the present moment. Often, the pressure to "perform" during sex can lead to anxiety, tension and less enjoyment. Sensate focus is about being in the moment and using your five senses (hearing, seeing, touching, listening and tasting) to help you and your partner focus on the sensations that are produced by exploring each other's bodies. These exercises start with an agreement for no genital contact, and gradually progress through a series of stages at a pace that feels comfortable for both partners.

Sensate focussing exercises are done in three stages. In order to get the maximum benefit, try to practice each stage 3 times per week for two or three weeks before advancing to the next stage – however, that is just a suggestion and you can do whatever feels best and right for you. Remember it is okay if you do not progress past the first stage, and if the first stage feels too much to start with it is okay to do adapt this, e.g. to start with doing this fully clothed or to specify parts of the body that you feel comfortable touching or being touched (e.g. just the hands or feet).

For detailed information about this exercise visit <a href="https://sexualwellbeingforall.files.wordpress.com/2019/07/sensate-focus-2019.pdf">https://sexualwellbeingforall.files.wordpress.com/2019/07/sensate-focus-2019.pdf</a>

Another way we can improve the conditions of sex is through psychological arousal and to do this we can use fantasies. Fantasies are internal images and stories which are very common for everyone to experience. Sexual fantasies can be used to help trigger sexual arousal. Often we cannot control sexual fantasies and it is common for violent fantasies to be experienced following sexual assault. This is not something you choose to experience, it is the way our brains process and codes our experiences. Even if you become aroused by an unwanted fantasy, it doesn't mean you enjoy/enjoyed it or want it - tricky brain can make associations that we don't necessarily want. This is termed arousal non-concordance when your brain is aroused by something you don't want. It is common and okay.

Just like the inner critic, we cannot force violent fantasies away but we can learn to develop new fantasies as our brains able to learn new skills. Some people may feel guilty about having unwanted fantasies but there is no such thing as wrong thoughts or feelings. What is more important is how you treat yourself when these difficulties arise. We can try be kinder to ourselves about the fantasies we have and reduce the shame associated with the fantasies

Sexual fantasies are normal and involves you trusting yourself and letting your imagination go.

With any of these practices, they may feel like a big step and that's understandable and okay, go at your own pace.

Returning to sex after trauma is understandably challenging and there is no reason to be critical or harsh with yourself if you're finding it more difficult. As we mentioned in the first session, your tricky brain sets off your threat system thinking it is protecting you. It is also an experience many survivors of sexual trauma experience, there is nothing wrong with you if you have any difficulties or no difficulties returning to sex. Over the last four sessions we hope we have deepened your understanding of your difficulties and through that understanding you have learnt to be more compassionate with yourself as your current experience is not your fault.

We hope that you have learnt some new skills as well to help you reduce the negative experience you may have during sex. We encourage you to continue practicing any of the exercises you found helpful throughout the four weeks. You will also be able to keep the handouts and refer back to them at any time.

We would like to thank you for attending each week and for continuing to fill in the measures. Your participation will aid future research into providing resources for survivors of sexual trauma with difficulties returning to sex. Thank you for taking part in this study, please fill in measures for the week. Afterwhich, we will be in touch with you in four weeks to check in on how you are doing.

## **Session 4: Handout**

## **Exercise: Compassionate Colour**

Reflections:

## Conditions for good sex



## Relationships

After traumatic sexual experiences, some people might notice a difference in their relationships or interactions with partner/s.

- Some partners may be understanding by responding with empathy and patience in relation to sexual intimacy
- Others may struggle to understand, and could take a less helpful stance

If you are currently with a sexual partner/s, or would like to enter into a romantic or sexual relationship in the future, it can be helpful to reflect on the dynamics between you and your partner/s and consider the following:

- How understood do you feel?
- How safe do you feel to engage in sex?
- How supportive is your partner of your needs and the pace you would like to take things?
- Are your 'conditions for enjoying sex and intimacy' being met?

## Activities involving physical touch

<u>Self Practice</u> or masturbation is another technique you can use to feel more in tune with your own body. It can help you regain some control over your body and understand more about what feels pleasureable for you.

For detailed information about this exercise:

 $\underline{https://sexualwellbeing for all.files.word press.com/2019/05/mindful-self-practice-for-those-with-a-vulva-1.pdf}$ 

<u>Sensate Focus</u> is a set of exercises geared towards couples where the focus of sex is shifted from pursuing orgasmic outcome, to a slower appreciation of physical intimacy and sensations. Removing the pressure to achieve orgasm allows the partners to connect more deeply within the present moment

For detailed information about this exercise:

https://sexualwellbeingforall.files.wordpress.com/2019/07/sensate-focus-2019.pdf

<u>Sexual Fantasies</u> are images and stories that trigger arousal and helpful in providing conditions for good sex. You can use fantasies to help with arousal and desire. However, it is also common for violent fantasies to be experience after sexual trauma. Even if you become aroused by an unwanted fantasy, it doesn't mean you enjoy/enjoyed it or want it - tricky brain can make associations that we don't necessarily want. Some people may feel guilty about having unwanted fantasies but there is no such thing as wrong thoughts or feelings. What is more important is how you treat yourself when these difficulties arise.

Using fantasies are a great way to elicit sexual arousal and is completely normal & natural healthy expression of your sexuality. Fantasies can be about whatever you want and you can use then during self practice or with a partner – try it if you are comfortable and if you aren't that's alright.

#### Week 4 Practice:

If you feel comfortable, try any or all of the exercises covered in this session throughout the week. There is no need to force yourself if you don't feel ready – you are in control and have the choice.

Thank you for engaging in these materials over the last 4 weeks. We hope you continue to practice being kind and compassionate with yourself even if you are still finding returning to sex difficult. That's okay. You took a big step to continue to engage in these materials and that is enough.

## **Appendix**

## Appendix A

#### **Signposting and Support Handout**

#### **Mental Health Support Lines:**

Samaritans – Offers free 24/7 support.

Call 116 123 or email jo@samaritans.org (24 hours, every day)

**SHOUT** – Offers free 24/7 mental health support text service if you prefer not to talk.

Text SHOUT to 85258 (24 hours, every day)

**Campaign Against Living Miserably (CALM)** – Offers our of hours support (5pm – midnight, everyday)

Call 0800 58 58 58 or their webchat service through the website

**SANEline** – Offers out of hours mental health support (4pm to 10pm everyday)

0300 304 7000

#### **Support related to sexual violence and abuse:**

Rape Crisis England & Wales - Provides information and support to survivors of sexual violence, sexual assault and sexual abuse across England and Wales.

Freephone 0808 802 9999 (12 to 2.30pm, then 7 to 9.30pm, every day) www.rapecrisis.org.uk

**Rape Crisis Scotland** - Provides information and support to survivors of sexual violence, sexual assault and sexual abuse across Scotland.

Freephone 0808 801 0302 (6pm to 12am, every day) www.rapecrisisscotland.org.uk

**Nexus NI** - Offers free counselling for people who have experienced sexual violence, sexual assault and sexual abuse across Northern Ireland. <a href="http://nexusni.org/">http://nexusni.org/</a>

**Galop** - Galop gives advice and support to people who have experienced biphobia, homophobia, transphobia, sexual violence or domestic abuse. They also support lesbian, gay, bi, trans and queer people who have had problems with the police or have questions about the criminal justice system.

Helpline: 020 7704 2040 http://www.galop.org.uk

National Association for People Abused in Childhood (NAPAC) - Offers support to adult survivors of childhood abuse.

Support line 0808 801 0331 (10am to 9pm, Monday to Thursday, and 10am to 6pm on Friday) <a href="https://napac.org.uk/">https://napac.org.uk/</a>

**Southall Black Sisters** - Campaigning, information and advice for women affected by gender-based violence.

Helpline: 0208 571 0800 http://www.southallblacksisters.org.uk/

**FORWARD** - Advice, support and specialist health care for girls and women affected by FGM. FORWARD is staffed by sensitive and approachable African women who as well as English speak Arabic and several other African languages.

Helpline: +44 (0)20 8960 4000 http://www.forwarduk.org.uk/resources/support

#### **Guided meditations for self-compassion:**

• <a href="http://self-compassion.org/category/exercises/#guided-meditations">http://self-compassion.org/category/exercises/#guided-meditations</a>

#### Mindfulness apps

- Headspace
- The Mindfulness App
- Mindfulness Daily
- ACT Coach
- Calm

Sexual pain: <a href="http://www.scarleteen.com/node/85">http://www.scarleteen.com/node/85</a>

A website dedicated to exploring the many ways that women can experience sexual pleasure. Includes videos and tutorials: www.omgves.com

#### Appendix B

## Communicating with a partner about level of comfort with sex after trauma

#### Ground Rules & Boundaries:

Ground rules should be established before the discussion to create an environment that allows partners to share their feelings in a safe way. It may be helpful to write these down to refer back to if needed. You may not agree on everything and that's okay, having ground rules ensures each view is expressed and respected.

Listening: Listening actively, trying to understand your partners point of view. Being emphatic and listening with your full heart. Understanding their difficulties, desire, feelings and action.

#### During this talk you can discuss with your partner

- → The impact of sexual trauma and how it affects the way survivors return to sex this is physiological and biological response that you have no control over and is not your fault. (You may choose to share or discuss the brains alarm system from session 1)
- → the level of comfort with sex are there any dos or don'ts specific to you? Anything you would prefer your partner to do/not do? This can start very simple e.g. holding hands, dancing, cuddling up in bed with a film. It can then branch into sexual things you feel comfortable with. You can compare ideas with your partner and see if anything on your 'safe' list also appeals to them.
- → Go through the sexual activities list and body map together
- → What sexual terms are off limits?
- → Agree to stay away from shaming each other
- → Be as specific as you can, giving examples of what you mean and offer different options for solutions with the understanding that these options can be negotiated and compromised on.
- → Tell your partner what they do well, not just what needs to be changed
- → Grounding techniques that you can use together
- → Safe words to use if either of you are feeling uncomfortable at any point and how that is not a sign of rejection but a pause to look after yourself.

## Appendix C

## **Sexual Activities List and Body Map**

Using the sexual activities list and/or body map as guidance to reflect on areas you are happy to explore with your partner or the areas you are less happy to explore.

You **do not** need to share this list with your partner, this list is for you to use. Share only what you are comfortable with.

| Anal Sex | Massage | You can include your own |
|-----------------|----------------------|--------------------------|
| Cuddling | Masturbation | activities as well |
| Cunnilingus | Sexting | |
| Ejaculation | Sex Toys | |
| Eye Contact | Slapping (where) | |
| Face Sitting | Phone Sex | |
| Fellatio | Teasing | |
| Foot Play | Tickling (where) | |
| Fingering | Touching (where) | |
| Hand Holding | Vaginal Pentetration | |
| Handjob | Watching | |
| Hair Pulling | 69 | |
| Kissing (where) | | |
| Lingerie | | |

# Looking at the images below, reflect on what areas you are happy to explore and which areas you are not ready to.

This activity can be done on your own before discussion with a partner if you feel ready to do so.. You do not need to share the body map with them if you are not comfortable



#### Appendix E

Compassionate Letter Writing developed by Paul Gilbert

The purpose of compassionate letter writing is to help you **refocus your thoughts and feelings on being supportive, helpful and caring of yourself**. In *practicing* doing this it can help you access an aspect of yourself that can help tone down negative feelings and thoughts.

The key of this exercise is to **practice becoming inwardly gentle, kind, compassionate and self supportive**. It takes time to build this compassionate muscle. You can practice thinking about how, each day, you can become more and more as you wish to be. As in all things there will be good times and not so good. Spend time imagining your postures and facial expressions, thoughts and feelings that go with being compassionate and practice creating these inside you. This means being open with our difficulties and distress, rather than just trying to get rid of them.

To start your letter, try to feel that part of you that can be kind and understanding of others; how you would be if caring for someone you liked. Draw upon the qualities you would like your compassionate self to embody. You do not have to feel like is who you are currently to draw on being compassionate.

As you write your letter, try to allow yourself to have *understanding and acceptance* for your difficulties and distress. For example, your letter might start with "I am sad you feel distressed; your distress is understandable because......" Note the reasons; realizing your distress makes sense. Then perhaps you could continue your letter with... "I would like you to know that......" (e.g., your letter might point out that as we become depressed, our depression can come with a powerful set of thoughts and feelings – so how you see things right now may be the depression view on things).

You can consider the following when writing your letter but you do not need to cover them all. Alternatively, you can write different things in different letters to yourself. As you write these letters avoid telling yourself what you should or should not think, feel or do. There is no right ot wrong, it is the process of trying to think in a different way that is important

Standing Back: Once you have acknowledged your distress and not blamed yourself for it, it is useful if your letter can help you stand back from the distress of your situation for a moment. If you could do that, what would be helpful for you to focus on and attend to?

*Not alone*: When we feel distressed we can often feel that we are different in some way. However, rather than feeling alone and ashamed remember many others can feel depressed with negative thoughts about themselves, the world or their future.

Reduce Self criticism: If you are feeling down, disappointed or are being harsh on yourself, note in your letter that self criticism is often triggered by disappointment, loss or fear. So we need to acknowledge and be understanding and compassionate about the disappointment, loss or fear. Allow yourself to be sensitive to those feelings.

Compassionate behavior: It is useful to think about what might be the compassionate thing to do at this moment or at some time ahead – how might your compassionate part help you do those things? So in your letter you may want to think about how you can bring compassion into action in your life. If there are things you are avoiding or finding difficult to do, write down some small steps to move you forward. Try to write down steps and ideas that encourage you and support you to do the things that you might find difficult.

*Dilemmas:* If you are in a dilemma about something, focus on the gentle compassionate voice inside you and write down the different sides of the dilemma. Note that dilemmas are often difficult, and at times there are hard choices to be made. Therefore, these may take time to work through. Talking through with others might be a helpful thing to do. Acceptance of the benefits and losses of a decision can take time.

Compassion for feelings: Your compassionate side will have compassion for your feelings. If you are having powerful feelings of frustration, anger or anxiety, then compassionately recognize these. Negative emotions are part of being human and can become more powerful in depression or when we are distressed but they do not make you a bad person – just a human being trying to cope with difficult feelings. Your compassionate mind will remind you that we often don't choose to feel negatively and these feelings can come quite quickly. In this sense it is 'not our fault', although we can learn how to work with these difficult feelings and take responsibility.

What is helpful: Your letter will be a way of practicing how to really focus on things that you feel help you. If thoughts come to mind that make you feel worse, then notice them, let them go and refocus on what might be helpful – remember there are no 'I shoulds'.

*Warmth:* Now try to focus of the feelings of warmth and genuine wish to help in the letter as you write it. Spend time breathing gently and really try, as best you can, to let feelings of warmth be there for you. When you have written your letter, read it through slowly, with as much warmth as you can muster. If you were writing to somebody else would you feel your letter is kin.

Remember that this is an exercise that might seem difficult to do at times but with practice you are exercising a part of your mind that can be developed to be helpful to you. Some people find that they can rework their letters the next day so they can think through things in a different way. The key of this exercise is the desire and effort of becoming inwardly gentle, compassionate and self-supportive. The benefits of this work may not be immediate but like 'exercising to get fit' can emerge over time with continued practice. Sometimes people find that even though they are depressed they would very much like to develop a sense of self that can be wise and compassionate to both themselves and others. You can practice thinking about how, each day, you can become more and more as you wish to be. As in all things there will be good times and not so good. Spend time imagining your postures and facial expressions, thoughts and feelings that go with being compassionate and practice creating these inside you.

This means being open with our difficulties and distress, rather than just trying to get rid of them.

Exercise by Paul Gilbert (2007)

## Additional optional activity: building on the sensual self

If you would like to add an additional component to the compassionate letter, it is encouraged that you reflect on how you would like to build on your sensual self and also write this down in the letter. What kind of activities can you do for yourself that is for no one else. What makes you feel good about yourself? How would you like your sensual self to feel? You can incorporate aspects of compassion here as well. There is no need to be harsh or critical with yourself here but hold yourself with nurturing compassion.